CLINICAL TRIAL: NCT00701077
Title: DAPERB 3,4-DiAminoPyridine and Electrophysiological Response in Brugada Syndrome
Acronym: DAPREB
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: recruitments issues
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P060802; EUDRACT 2007-004133-42
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Brugada Syndrome
Keywords: Brugada syndrome; Electrophysiological study; Ion channel blockade
MeSH Terms: conditions — Brugada Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 3,4-Di-amino-Pyridine : a single 20 mg dosing
  Interventions: Drug: 3,4-Di-amino-Pyridine
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 3,4-Di-amino-Pyridine — a single 20 mg dosing
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
The Brugada syndrome is a rare disease potentially leading to severe arrhythmic events in otherwise healthy subjects.In many patients an Implantable cardiovertor defibrillator (ICD) is implanted to prevent sudden cardiac death. ICD are however associated with potential complications and are not available in all countries.Pharmacological blockade of specific ion channels (Ito) represents a promising therapeutic approach in this syndrome.The 3,4-diaminopyridine (3,4-DAP) is a pharmacological Ito blocker that can be used in humans.The aim of the study is to evaluate the effect of 3,4-DAP on ventricular arrhythmia inducibility in Brugada patients requiring an electrophysiological study for arrhythmic risk stratification.

DETAILED DESCRIPTION:
Background:

The Brugada syndrome is a rare disease potentially leading to severe arrhythmic events in otherwise healthy subjects.In many patients an Implantable cardiovertor defibrillator (ICD) is implanted to prevent sudden cardiac death. ICD are however associated with potential complications and are not available in all countries.Pharmacological blockade of specific ion channels (Ito) represents a promising therapeutic approach in this syndrome. Experimental data show that increased Ito current may be associated with both the ECG feature and arrhythmogenic substrate observed in the syndrome. Moreover, Ito blockade reverse the ECG abnormalities and suppress arrhythmogenicity.The 3,4-diaminopyridine (3,4-DAP) is a pharmacological Ito blocker that is already used in humans for another indication.

Main objective:

The aim of the study is to evaluate the effect of 3,4-DAP on ventricular arrhythmia inducibility in Brugada patients requiring an electrophysiological study for arrhythmic risk stratification.

First end point:

Re-inducibility or non re-inducibility of sustained ventricular arrhythmia during electrophysiological study on treatment

Tested hypothesis:

The 3,4-DAP decreases the proportion of re-inducibility during the electrophysiological study with a re-inducibility rate of 80% in the placebo group and 25% in the 3,4-DAP group

Secondary objective:

* to assess the effect of 3,4-DAP on ST segment elevation in Brugada patients
* to describe the relationship between 3,4-DAP plasma concentration measured at 45 minutes and electrophysiological study result and ST segment elevation

Study design:

2 centres, randomised, double blind, parallel groups, placebo controlledA single dose of 20 mg of 3,4-DAP

Included patients and number of patients:

Included patients will all have a diagnosed Brugada type 1 ECG and will require an electrophysiological study for arrhythmic risk stratification purpose. Only inducible patients will be included in the study.Using a classical approach, the hypothesis would be that 80% of on placebo patients would be re-inducible when only 25% of on drug patients would. To test such an hypothesis, 32 patients (16 in each group) would have been necessary (a=5%, b=20%).Provided the essential binary response of the electrophysiological study we choose a sequential approach in order to get the opportunity stop for success or futility the inclusions before the end of the study. The maximum number of included patients will then be 42 (21 in each group).

Protocol duration:

Study duration is 48 hours for each patient.The protocol duration is planned for 5 years.

Per protocol procedures:

* Electrophysiological study with ventricular programmed stimulation performed twice
* Continuous ECG recording- Blood sampling for 3,4-DAP plasma concentration measurement Potential implications:If the study hypotheses are confirmed it would then be justified to design long term efficacy studies in Brugada patients implanted with an ICD.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman ≥ 18 years old
* Brugada syndrome diagnosed with a type 1 ECG either spontaneous or drug-induced
* Electrophysiological study indicated for arrhythmic risk stratification purpose
* Inducibility of a sustained ventricular tachycardia (> 30 seconds) or ventricular fibrillation requiring defibrillation
* Physical medical examination
* Signed written informed consent

Exclusion Criteria:

* Personal or familial history of epilepsy
* Pregnancy
* Body weight > 100 kg
* the need of >1 counter shock for defibrillation
* Alcohol or cocaine consumption during the protocol
* Class I (with the exception of local anaesthesia by lidocaine), II, III and IV antiarrhythmic drugs, antidepressant drugs, ATP dependent potassium channel activators, sultopride not stopped for > 7 halve-lives
* No medical insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-09-12 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Electrophysiological study result (re-inducibility or not) 45 minutes after drug intake | 45 minutes after drug intake

SECONDARY OUTCOMES:
the effect of 3,4-DAP on ST segment elevation in Brugada patients (45 minutes) | at 45 minutes
the relationship between 3,4-DAP plasma concentration measured at 45 minutes and electrophysiological study result and ST segment elevation | at 45 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice EXTRAMIANA, MD, PhD, Principal Investigator — Lariboisière University Hospital - Cardiology Department
Locations (1):
- Lariboisière University Hospital - Cardiology department, Paris, France